CLINICAL TRIAL: NCT00601393
Title: Interactive Internet Intervention for Depressed Mothers
Brief Title: Effectiveness of Internet-Based Cognitive Behavioral Therapy for Treating Mothers With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH070426 (NIH); R01MH070426 (NIH); DSIR CT-C
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants will receive treatment as usual followed by 8 weeks of Internet-based cognitive behavioral therapy treatment
  Interventions: Behavioral: Cognitive behavioral therapy (CBT); Other: Treatment as usual (TAU)
- 2 (Experimental): Participants will receive 8 weeks of Internet-based cognitive behavioral therapy treatment
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — CBT treatment is delivered via the Internet. Adaptations to the CBT program will include the addition of content of particular relevance to mothers of young children and the incorporation of instructional design principles to promote self-learning. The treatment program will take advantage of the unique properties of the Internet, including multimedia presentations and interactive components with professional and moderated peer social support.
Other: Treatment as usual (TAU) — Participants receiving TAU will be offered the CBT treatment after a wait-list period. During the wait-list period, participants will be offered facilitated referrals to treatment provided in the community.
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of an Internet-based cognitive behavioral therapy program in treating mothers with depression who have young children.

DETAILED DESCRIPTION:
Being a mother of a young child can be very stressful. Many women find that being a parent may not be as enjoyable as expected and that they feel persistently tired or sad. Because of the possible "lows" of recent motherhood, new mothers are particularly prone to depression. The impact of depression on recent mothers is significant, including emotional distress for the woman as well as possible disturbances in the child's development. If left untreated, the mother's depression may cause strain on family life and her relationship with her child. Cognitive behavioral therapy (CBT), a form of psychotherapy that can be used to treat people with depression, aims to modify thoughts and behaviors. Despite the availability of helpful CBT programs, most depressed people do not receive treatment. To make these treatments more accessible to mothers who may lack the means to seek help, this study will adapt CBT for depression to an at-home computer-based program. This study will evaluate the effectiveness of the computer-based CBT program in improving the moods of depressed mothers and their children and enhancing the quality of time shared between mother and child.

Participation in this single-blind study will last at least 8 weeks. A computer, modem, monitor, and Internet connection will be installed in the homes of all participants. Participants will then be randomly assigned to receive either immediate treatment or delayed treatment, which will begin after a wait-list period. Treatment will be delivered on a computer, which will allow the participants to chat online with other parents and their program coach. There will be 11 CBT-related lessons over 8 weeks, taking between 8 and 11 hours total to complete. The lessons will promote self-learning and will include content of particular relevance to mothers of young children, including how to handle stress and improve mood. Participants will be required to contact their coach at least every 2 weeks to review the lessons learned. There will be three assessments, occurring at pretreatment, immediately post-treatment, and 3 months post-treatment. Participants assigned to delayed treatment will complete one additional assessment prior to beginning the wait-list period. Each assessment will involve both parent and child and will include play interactions, questionnaires, and interviews about parenting, feelings, child behavior, moods, and self-esteem. Another caretaker of the child and the child's teacher will also be asked to complete questionnaires about the child's and/or parent's behavior.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of elevated self-reported depressive symptomatology, confirmed by a CES-D score of greater than 21
* Understands spoken English
* Either the biological/adoptive mother, permanent legal guardian, or long-term relative caretaker for the child
* Resides in a stable residence with the infrastructure for phone service that can support Internet access

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies-Depression (CES-D) Scale | Measured at pretreatment, post-treatment, and 3-month follow-up

SECONDARY OUTCOMES:
Dyadic Parent Child Interaction Coding System | Measured at pretreatment, post-treatment, and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lisa B. Sheeber, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Sheeber LB, Seeley JR, Feil EG, Davis B, Sorensen E, Kosty DB, Lewinsohn PM. Development and pilot evaluation of an Internet-facilitated cognitive-behavioral intervention for maternal depression. J Consult Clin Psychol. 2012 Oct;80(5):739-749. doi: 10.1037/a0028820. Epub 2012 Jun 4. PMID 22663903